CLINICAL TRIAL: NCT02107248
Title: The Need for Supine Position Advise During Sleep in the First 8 Week After a Total Hip Replacement to Prevent Hip Dislocation
Brief Title: Supine Sleeping After Total Hip Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orthopedisch Centrum Oost Nederland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL4670604413; P13-31 METC Twente (Registry Identifier: Medical Ethical Committee Twente)
Record Dates: First submitted 2014-04-03; First posted 2014-04-08 (Estimated); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Osteoarthritis; Hip Dislocation
Keywords: Arthroplasty; Replacement; Hip; Posterolateral surgery; Precautions
MeSH Terms: conditions — Osteoarthritis; Hip Dislocation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sleep position: supine (Active Comparator): Subjects will be instructed to sleep in a supine position during the first eight weeks after a total hip replacement following a posterolateral surgical approach
  Interventions: Behavioral: Sleep position: supine
- Sleep position: no restrictions (Experimental): Patients do not have any restrictions in sleeping position during the first eight weeks after a total hip replacement following a posterolateral surgical approach
  Interventions: Behavioral: Sleep position: no restrictions

INTERVENTIONS:
Behavioral: Sleep position: no restrictions — during the first eight weeks after total hip replacement following a posterolateral surgical approach
  Arms: Sleep position: no restrictions
Behavioral: Sleep position: supine — during the first eight weeks after total hip replacement following a posterolateral surgical approach
  Arms: Sleep position: supine

SUMMARY:
Aim of the current study is to test the non-inferiority hypothesis of differences in early hip dislocation between a group of patients who will be restricted to sleep in supine position and a group without restricted sleeping position during the first eight weeks after a total hip replacement following a posterolateral surgical approach

DETAILED DESCRIPTION:
stratified block randomized controlled trial

ELIGIBILITY:
Inclusion Criteria:

* Placement of a primary total hip replacement via the posterolateral approach by a high volume orthopaedic surgeon
* Patients with a ASA-classification of I or II

Exclusion Criteria:

* Blindness
* Replacement of 2nd total hip within six months after the1st total hip replacement surgery
* Insufficient knowledge of the Dutch language
* Collum fracture
* Infection of total hip replacement
* Cognitive dysfunction
* Wheelchair dependability
* Hypermobility
* Alcohol abuse
* Neurological disorders such as Parkinson and stroke

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 456 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Percentage early hip dislocations | in first eight weeks after THP

SECONDARY OUTCOMES:
HOOS | eight weeks and six months post-operative
  Hip Disability and Osteoarthritis Outcome Score
VHS | eight weeks and six months post-operative
  Quality of Sleep
EQ-5D | eight weeks and six months post-operative
  Quality of Life
VAS/NRS hip | eight weeks and six months post-operative
  pain intensity
Compliance anti-dislocation instructions | eight weeks post-operative
  diary for patients to report their compliance with the set of anti-dislocation instructions, among which is the (daily) reporting of their sleeping position in bed at night

OTHER OUTCOMES:
Sleeping position preference | baseline
  necessary information for the stratification procedure

CONTACTS AND LOCATIONS:
Overall Officials: Anil Peters, Principal Investigator — Orthopedisch Centrum Oost Nederland
Locations (1):
- Orthopedisch Centrum Oost Nederland, Hengelo, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Peters A, Manning F, Tijink M, Vollenbroek-Hutten M, Huis In 't Veld R. Patient compliance with postoperative precautions in an unrestricted and a supine sleeping position following posterolateral total hip arthroplasty: a randomized controlled trial. Disabil Rehabil. 2022 Dec;44(26):8303-8310. doi: 10.1080/09638288.2021.2012606. Epub 2021 Dec 21. PMID 34932433
- [Derived] Peters A, Tijink M, Veldhuijzen A, Huis in 't Veld R. Reduced patient restrictions following total hip arthroplasty: study protocol for a randomized controlled trial. Trials. 2015 Aug 18;16:360. doi: 10.1186/s13063-015-0901-0. PMID 26283079